CLINICAL TRIAL: NCT00274417
Title: A Randomized, Placebo-Controlled, Double-Blind Study of the Use of Dutasteride for Improving Peri-Operative and Long-Term Outcomes of Photoselective Vaporization of the Prostate (DOP Study)
Brief Title: Dutasteride for Improving Peri-Operative and Long-Term Outcomes of Photoselective Vaporization of the Prostate (DOP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Urology of Virginia (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UVA-001
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-04

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Dutasteride

INTERVENTIONS:
Drug: dutasteride

SUMMARY:
This study is for individuals electing to have GreenLight Photoselective Vaporization of the Prostate (PVP) to treat symptoms from an enlarged prostate gland. The purpose of this research study is to evaluate the safety and effectiveness of the medication dutasteride as compared to placebo (an inactive substance) for improving surgical and long-term outcomes of PVP. Dutasteride is approved by the United States Food and Drug Administration (FDA) for the treatment of symptoms from an enlarged prostate gland. The use of dutasteride to improve the outcomes of PVP is investigational. The study will last for approximately 15 months and will involve 6 visits.

DETAILED DESCRIPTION:
The purpose of the study is to assess the effects of dutasteride on the outcomes and QoL of patients undergoing GreenLight Photoselective Vaporization of the Prostate. PVP is a growing, outpatient surgical treatment for BPH. The addition of dutasteride may potentially improve both the short and long term outcomes. Use peri-operatively may improve visibility during surgery, shorten operative time, lessen bleeding both intra and post-operatively and hasten post-op recovery. Continued use long-term (12 months following the procedure) may improve overall symptomatic scores as combination therapy with PVP. The addition of dutasteride to PVP may decrease the occasional occurrence of continued post-op irritative symptoms and lessen the likelihood of the need for re-catheterization with overall improvement in quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged ≥ 50 years old 2. Subjects with LUTS due to BPH with:

1. AUA SI score ≥ 12 at baseline
2. Qmax ≤ 15 mL/sec (on at least 125 mL)
3. Symptoms for ≥ 3 months 3. Subjects with prostate volume ≥ 30 grams 4. Subjects who are appropriate surgical candidates for Photoselective Vaporization of the Prostate (PVP) as determined by a study investigator 5. Subjects able to swallow and retain oral medication 6. Subjects able to comply with study protocol 7. Subjects able to read and write (to complete the self-administered AUA SI) 8. Subjects who sign the approved Informed Consent Form for the study

   Exclusion Criteria:
   1. Subjects who have previously undergone a surgical treatment for BPH including but not limited to TURP, TUNA, TUIP, thermotherapy, prostatic stent, dilation balloon, etc.
   2. Subjects with a history of prostate cancer
   3. Subjects with a history of bladder or testicular cancer in the past 5 years

       Subjects who have been cancer-free for at least 5 years will be eligible

       Subjects with a history of superficial bladder cancer will not be excluded
   4. Subjects who have received radiation to the pelvis or prostate or radical surgery to the pelvic area
   5. Subjects with persistent gross hematuria, current symptomatic prostatitis
   6. Subjects with neurogenic bladder and/or sphincter abnormalities for any reason including Parkinson's disease, multiple sclerosis, stroke, or diabetes
   7. Subjects who have used any 5 α-reductase inhibitors in the past 3 months.

       Subjects who wash-out of these medications for 3 months prior to screening will be eligible
   8. Subjects taking alpha-blockers within 2 weeks prior to randomization.

       Subjects must be off of alpha blockers at the time of randomization for the measurement of AUA Symptom Score, QoL Score, flow rate, post void residual, etc. In the rare case a patient goes into retention during the 3 month period between randomization and PVP, they will be allowed to resume their alpha blocker until the PVP since no outcomes are measured during this period. They will be required to discontinue the alpha blocker after they have surgery
   9. Subjects on an unstable regimen of antidepressants, anticholinergics, androgens, or herbal supplements including phyto-sterols (such as saw palmetto)  Subjects who are on a stable regimen of the above medications for at least 1 month prior to screening and are willing to stay on the same dose for the duration of the study will be eligible
   10. Subjects on an unstable regimen of beta-blockers, antihistamines, anticonvulsants, antispasmodics, or other medications known to affect the clinical symptoms of BPH

        Subjects who are on a stable regimen of the above medications for at least 4 months prior to screening and are willing to stay on the same dose for the duration of the study will be eligible
   11. Subjects with a post void residual > 350 mL
   12. Subjects with a known hypersensitivity to 5α-reductase inhibitors
   13. PSA > 10  Subjects with a PSA between 4 and 10 with a negative prostate biopsy and deemed at low risk for prostate cancer by the investigator
   14. Subjects with serum creatinine >1.5 x the upper limit, ALT > 2 x the upper limit, AST > 2 x the upper limit, ALP > 2 x the upper limit, or bilirubin > 1.5 x the upper limit for normal
   15. Subjects treated in the last 30 days with another investigational product or currently participating in another study with an investigational drug or procedure
   16. Subjects deemed ineligible for the study by the site investigators or the sponsor

       -

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2006-01; Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Change in American Urologic Association Sympton Score

SECONDARY OUTCOMES:
Change in BPH Quality of Life
Change in urinary flow rate
Change in post void residual
PVP operation time, wattage use, estimated blood loss
Post-operative catheter time
Incidence of post-operative dysuria and hematuria
Incidence of expected and unexpected adverse events following PVP

CONTACTS AND LOCATIONS:
Overall Officials: Gregg Eure, MD, Principal Investigator — Urology of Virginia Research, Devine-Tidewater Urology
Locations (2):
- United States (2):
  - Urology of Virginia, Norfolk, Virginia
  - Urology of Virginia, Virginia Beach, Virginia